CLINICAL TRIAL: NCT07031960
Title: Design, Construction and Evaluation of the Educational Effects of 3D Simulator of Human Eyeball Movements
Brief Title: 3D Eye Movement Simulator for Medical Education
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, mehrnoush malekzadeh, Assistant Professor, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IR.ARI.MUI.REC.1404.051
Record Dates: First submitted 2025-06-09; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Education; Education, Medical, Undergraduate; Education, Medical
Keywords: medical education; 3D model; eye movement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D Eyeball Movement Simulator Group (Experimental): Arm 1 (Experimental Group): Participants in this arm will use an interactive 3D-printed simulator that physically replicates human eyeball movements and extraocular muscle function. This hands-on educational tool allows medical students to manipulate the model and observe biomechanical principles of eye movements in real-time.
  Interventions: Device: 3D Eyeball Movement Simulator Group
- Conventional Teaching Methods Group (Active Comparator): Participants in this arm will receive standard anatomy instruction through traditional methods including didactic lectures, 2D textbook illustrations, and static anatomical models - representing the current typical curriculum for ophthalmic anatomy education.
  Interventions: Other: Conventional Teaching Methods Group

INTERVENTIONS:
Device: 3D Eyeball Movement Simulator Group — A physical, interactive 3D-printed educational model that replicates human eyeball movements and demonstrates the biomechanical action of extraocular muscles. The simulator allows hands-on manipulation to demonstrate all cardinal eye movements (adduction, abduction, elevation, depression, intorsion, and extorsion) through mechanical actuation of synthetic muscle analogues."
  Arms: 3D Eyeball Movement Simulator Group
Other: Conventional Teaching Methods Group — Standard medical education methods for teaching eye anatomy and movements, including: (1) didactic classroom lectures with 2D illustrations, (2) static anatomical models of the orbit and eyeball, and (3) textbook-based learning materials. This represents the current conventional approach to teaching this content in medical curricula
  Arms: Conventional Teaching Methods Group

SUMMARY:
The goal of this clinical trial is to evaluate whether a new 3D-printed eyeball movement simulator improves medical education compared to traditional teaching methods. The main questions it aims to answer are:

Does using the 3D simulator help medical students better understand eye anatomy and muscle function compared to standard lectures and textbooks?

How do students rate the usability and effectiveness of this new teaching tool?

Researchers will compare two groups of medical students:

One group will learn using the 3D simulator

The other group will receive standard teaching methods

Participants will:

1. Complete a pre-test to assess their baseline knowledge
2. Attend training sessions using either the 3D simulator or standard methods
3. Take a post-test to measure learning improvement
4. Provide feedback about their learning experience
5. Take a post-intervention exam and satisfaction survey
6. Participate in focus groups about their learning experience

The study will help determine if interactive 3D models can enhance medical education about eye movements.

ELIGIBILITY:
Inclusion Criteria:

1. Academic Status Currently enrolled medical students in their preclinical years (typically 2nd-3 year)"
2. Course Enrollment "Formally registered in the special scence/anatomy course where eye movement education is part of the curriculum"

Prior Experience "No previous formal training in extraocular muscle anatomy or eye movement assessment"

Language Proficiency "Fluent in the language of instruction (Farsi)"

Consent "Willing and able to provide informed consent"

Exclusion Criteria:

1- Prior Exposure "Medical students who have previously taken advanced special scence courses"

Professional Experience "Students with prior clinical experience in ophthalmology ( as nurses or technicians)"

Atypical Curriculum "Students from schools with non-standard anatomy curricula that already include similar 3D simulation tools"

Participation Conflicts "Currently participating in other educational research studies that could confound results"

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Knowledge Gain Score | Baseline (pre-intervention), Immediately after intervention (1 day post-training)
  Difference in test scores between pre-intervention and post-intervention assessments on eye anatomy and movement kinematics, measured using a validated 50-point multiple-choice questionnaire

SECONDARY OUTCOMES:
Skill Acquisition in Eye Movement Assessment | "Baseline" or "Day 1"
  Performance in practical examination where students identify and demonstrate eye movements on standardized patients, scored by blinded evaluators using a 12-point checklist.
Student Satisfaction Scores | Immediately post-intervention
  Participant-reported satisfaction with the teaching method measured via 5-point Likert scale survey (1=very dissatisfied to 5=very satisfied).

IPD SHARING:
Plan to Share IPD: No